CLINICAL TRIAL: NCT03005158
Title: High-Sensitivity Cardiac Troponin On Presentation to Rule Out Myocardial Infarction (HiSTORIC): A Stepped Wedge Cluster Randomized Trial
Brief Title: High-Sensitivity Cardiac Troponin On Presentation to Rule Out Myocardial Infarction
Acronym: HiSTORIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PG/15/51/31596
Record Dates: First submitted 2016-08-15; First posted 2016-12-29 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: High-sensitivity cardiac troponin I; Myocardial infarction; Acute coronary syndrome; Cluster-randomized trial
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Validation Phase (Other): All six hospital sites currently use the ARCHITECT STAT high- sensitive troponin I assay in the assessment of patients with suspected acute coronary syndrome and use sex-specific thresholds upper reference limits (99th centile) to rule out myocardial infarction. This validation phase of up to 10 months will provide baseline information for each site on patients with suspected acute coronary syndrome in whom myocardial infarction is ruled out.
  Interventions: Other: Validation Phase
- Randomization Phase (Other): Participating centres will be randomized to implement the HighSTEACS pathway (intervention). The order of implementation will be randomized, with paired participating centres implementing in steps over a 6 month period.
  Interventions: Other: Randomization Phase
- Implementation Phase (Active Comparator): A final phase of up to 10 months after implementation of the HighSTEACS pathway will be matched by calendar month in each site to that of the validation phase, allowing each participating centre to act as its own control and to adjust for seasonal differences in the incidence of myocardial infarction and mortality.
  Interventions: Other: Implementation Phase

INTERVENTIONS:
Other: Validation Phase — Standard care across all sites during the validation phase will rule out myocardial infarction in those with presentation troponin below the 99th centile with greater than 6 hours of symptoms at the time of blood sampling. In those with less than 6 hours of symptoms, a second test will be measured 6- 12 hours after presentation.
  Arms: Validation Phase
Other: Randomization Phase — Standard care or HighSTEACS pathway.
  Arms: Randomization Phase
Other: Implementation Phase — Implementation of the HighSTEACS pathway to rule out myocardial infarction in patients with suspected acute coronary syndrome. Myocardial infarction will be ruled out if presentation cardiac troponin concentrations are <5 ng/L in those with at least 2 hours of symptoms at the time of blood sampling. In patients with less than two hours of symptoms, or where cardiac troponin concentrations are between 5ng/L and the 99th centile, repeat testing will be recommended at 3 hours. Myocardial infarction will be ruled out at 3 hours if cardiac troponin concentrations are unchanged (<3 ng/L change) and remain ≤99th centile on retesting. Those remaining ≤99th centile on retesting but demonstrating a significant change will require admission for further testing at 6-12 hours.
  Arms: Implementation Phase

SUMMARY:
Patients with suspected acute coronary syndrome account for a tenth of all presentations to the Emergency Department and up to 40 per cent of unplanned hospital admissions. The majority of patients do not have a heart attack (myocardial infarction), and may be safely discharged from the Emergency Department.

The investigators propose to evaluate whether the use of the HighSTEACS pathway in patients with suspected acute coronary syndrome reduces length of stay and allows more patients to be safely discharged from the Emergency Department. This pathways utilizes high-sensitivity cardiac troponin I testing and will rule out myocardial infarction if troponin concentrations are <5 ng/L on presentation, with further testing indicated at 3 hours only in those presenting early or with troponin concentrations between 5 ng/L and the 99th centile.

In six secondary and tertiary centres across Scotland, the investigators will introduce the pathway as part of a stepped wedge cluster randomized controlled trial. Sequential hypothesis testing will evaluate the efficacy and safety of the pathway. The primary efficacy end-point will be length of stay from time of presentation until final hospital discharge and the primary safety end-point will be survival free from type 1 or 4b myocardial infarction or cardiac death from discharge to 30 days. The study population will consist of those patients with cardiac troponin concentrations within the normal reference range (<99th centile) at presentation.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with suspected acute coronary syndrome
* High-sensitivity cardiac troponin I measured as part of routine clinical care

Exclusion Criteria:

* Patients who are not resident in Scotland
* Patients with ST-segment elevation myocardial infarction
* Patients presenting to hospital in cardiac arrest
* Patients with presentation high-sensitivity cardiac troponin I concentrations greater than sex-specific 99th centile thresholds

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31492 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay (minutes) | Length of time from initial presentation to the Emergency Department until final discharge from hospital, an average of 24 hours.
  This time frame is unique to each patient
Type 1 or type 4b myocardial infarction or cardiac death after discharge and within 30 days of index admission | Hospital discharge to 30 days after initial presentation

SECONDARY OUTCOMES:
Proportion of patients discharged directly home from the Emergency Department | Presentation to discharge from hospital, an average of 24 hours.
  Time frame of initial hospital episode is unique to each patient
Type 1 or 4b Myocardial Infarction after hospital discharge (independently double adjudicated using all available clinical information) | Hospital discharge to 30 days and 1 year after initial presentation
  An adjudicated diagnosis of type 1 and type 4b myocardial infarction will be made in line with the universal definition of myocardial infarction, using all available clinical information.
Cardiac death after hospital discharge (independently double adjudicated using all available clinical information) | Hospital discharge to 30 days and 1 year after initial presentation
Cardiovascular death after hospital discharge (independently double adjudicated using all available clinical information) | Hospital discharge to 30 days and 1 year after initial presentation
All-cause death after hospital discharge | Hospital discharge to 30 days and 1 year after initial presentation
Unplanned coronary revascularisation after hospital discharge (from cardiac intervention databases and case note review) | Hospital discharge to 30 days and 1 year after initial presentation
  We will identify any patients who require unplanned percutaneous coronary intervention or coronary artery bypass grafting.
Proportion of patients re-attending the Emergency Department | Hospital discharge to 30 days and 1 year after initial presentation

OTHER OUTCOMES:
Pre-specified sub-group analyses of the primary outcome | length of hospital stay defined as the length of time from initial presentation to the Emergency Department until final discharge from hospital; safety follow-up time frame of 30 days and 1 year after hospital discharge
  We will evaluate if the effect of intervention is significantly stronger or weaker in pre-specified sub-groups by assessing the co-primary endpoints in those who present with cardiac troponin <5 ng/L (low risk group), and in the whole population across different ages (considering age as a continuous variable), by duration of symptoms (considered as a continuous variable), by gender, by those who have or do not have a pre-existing history of ischaemic heart disease, by those with a presentation electrocardiogram suggesting ischaemia, by the GRACE risk score (considered as a continuous variable), and by day of patient presentation (assessing differences in weekday/weekend or routine/out-of-hours presentation).
Cost-effectiveness analysis | 1 year
  Based on costs of investigation and management in the year after initial hospital presentation

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L Mills, MD, PhD, Principal Investigator — University of Edinburgh; Ian Ford, PhD, Study Chair — University of Glasgow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shah AS, Anand A, Sandoval Y, Lee KK, Smith SW, Adamson PD, Chapman AR, Langdon T, Sandeman D, Vaswani A, Strachan FE, Ferry A, Stirzaker AG, Reid A, Gray AJ, Collinson PO, McAllister DA, Apple FS, Newby DE, Mills NL; High-STEACS investigators. High-sensitivity cardiac troponin I at presentation in patients with suspected acute coronary syndrome: a cohort study. Lancet. 2015 Dec 19;386(10012):2481-8. doi: 10.1016/S0140-6736(15)00391-8. Epub 2015 Oct 8. PMID 26454362
- [Background] Shah ASV, Anand A, Chapman AR, Newby DE, Mills NL; High-STEACS Investigators. Measurement of cardiac troponin for exclusion of myocardial infarction - Authors' reply. Lancet. 2016 Jun 4;387(10035):2289-2291. doi: 10.1016/S0140-6736(16)30517-7. No abstract available. PMID 27302263
- [Derived] Li Z, Doudesis D, Bularga A, Wereski R, Taggart C, Lowry MTH, Chapman AR, Tuck C, Ferry AV, Gray A, Newby DE, Anand A, Lee KK, Mills NL; HiSTORIC Trial Investigators. Safety of Using Risk Stratification Along With High-Sensitivity Cardiac Troponin in the Emergency Department: A Secondary Analysis. J Am Coll Cardiol. 2025 Nov 11;86(19):1738-1748. doi: 10.1016/j.jacc.2025.08.059. PMID 41193094
- [Derived] Anand A, Lee KK, Chapman AR, Ferry AV, Adamson PD, Strachan FE, Berry C, Findlay I, Cruikshank A, Reid A, Collinson PO, Apple FS, McAllister DA, Maguire D, Fox KAA, Newby DE, Tuck C, Harkess R, Keerie C, Weir CJ, Parker RA, Gray A, Shah ASV, Mills NL; HiSTORIC Investigatorsdagger. High-Sensitivity Cardiac Troponin on Presentation to Rule Out Myocardial Infarction: A Stepped-Wedge Cluster Randomized Controlled Trial. Circulation. 2021 Jun 8;143(23):2214-2224. doi: 10.1161/CIRCULATIONAHA.120.052380. Epub 2021 Mar 23. PMID 33752439
- [Derived] Ferry AV, Strachan FE, Stewart SD, Marshall L, Lee KK, Anand A, Shah ASV, Chapman AR, Mills NL, Cunningham-Burley S. Exploring Patient Experience of Chest Pain Before and After Implementation of an Early Rule-Out Pathway for Myocardial Infarction: A Qualitative Study. Ann Emerg Med. 2020 Apr;75(4):502-513. doi: 10.1016/j.annemergmed.2019.11.012. Epub 2020 Jan 23. PMID 31983496